CLINICAL TRIAL: NCT05587036
Title: A Randomized, Triple-blind, Placebo-controlled Study on the Effect of Rifaximin on Psychobiological Functions in Healthy Men
Brief Title: Effects of Rifaximin on Gut Microbiota and Emotion
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lukas Van Oudenhove, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: S66407; 2021-006814-35 (EudraCT Number)
Record Dates: First submitted 2022-09-29; First posted 2022-10-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers; Stress; Fear
Keywords: Rifaximin; Anti-Bacterial Agents; Stress; Fear; Inflammation; Short-Chain Fatty Acid; Microbiota-Gut-Brain Axis
MeSH Terms: conditions — Inflammation | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and personnel involved in data analyses are blinded to the intervention. Unblinding occurs after all data has been collected and analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rifaximin (Experimental): Rifaximin oral tablets, 550 mg, twice daily, two-weeks
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Placebo oral tablets, twice daily, two-weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin oral tablet, 550 mg, twice daily, two-weeks
  Other Names: Targaxan
  Arms: Rifaximin
Dietary Supplement: Placebo — Placebo oral tablet, twice daily, two-weeks
  Arms: Placebo

SUMMARY:
A randomized, triple-blind, placebo-controlled study on the effect of rifaximin on psychobiological functions in healthy men.

DETAILED DESCRIPTION:
This study is a randomized, triple-blind, placebo-controlled, interventional trial aiming to elucidate the impact of rifaximin-induced gut microbiota alteration to the psychobiological functioning of healthy men. The intervention will be performed in a parallel group design where one group will receive rifaximin (Targaxan 550 mg) twice daily for two weeks (treatment arm), while the other group will receive placebo (placebo arm).

Primary objective: to test the effect of rifaximin on stress sensitivity and fear-related processes

Secondary objective: to determine the mediating and/or moderating factors that underlie rifaximin-induced psychobiological changes

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Proficiency in English and/or Dutch
3. Healthy with no intestinal and/or psychological complaints
4. Access to a -18°C freezer (i.e. ordinary household freezer)
5. Male participants
6. Age 18-50 years
7. BMI 18.5-25 kg/m2

Exclusion Criteria:

1. Participant has a history of previous or current neurological, psychiatric, gastrointestinal or endocrine disorder
2. Any disorder, which in the Investigator's opinion might jeopardize the participant's safety or compliance with the protocol
3. Any prior or concomitant treatment(s) that might jeopardize the participant's safety or that would compromise the integrity of the Trial
4. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
5. Hypersensitivity to the active substance rifaximin, to any rifamycin (e.g. rifampicin or rifabutin) or any of the excipients
6. Current or recent medication use
7. Use of antibiotics within three months preceding the study
8. Current or recent (1-month) infection (e.g. common cold, influenza, COVID-19, etc.)
9. Previous or current substance/alcohol dependence or abuse (>2 units per day or 14 units per week)
10. One or more diagnoses based on the mini international neuropsychiatric interview (MINI-S)
11. One or more diagnoses based on ROME IV for gastrointestinal disorders
12. Smoking
13. Night-shift work
14. Adherence to special diets (e.g. vegan, vegetarian, weight-loss, lactose-free, gluten-free, etc.)
15. Use of pre- or probiotics within one month preceding the study
16. Previous experience with any of the tasks used in the study (not including questionnaires)
17. Color vision deficiency (colorblindness)
18. Magnetic Resonance Imaging (MRI) contraindications, including claustrophobia, severe back problems, conditions that would interfere with MRI scanning (e.g. cochlear implant, metal fragments in eyes, metallic body inclusion, or other metal implanted in the body), and if the participant does not want to be informed of incidental findings that might be found during imaging.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Stress sensitivity (biological) | Throughout study completion, on average 1 year
  Biological stress sensitivity is measured by quantifying cortisol levels (ng/ml) from multiple saliva samples taken before, during, and after a stress task performed during the pre-intervention and post-intervention visit.
Stress sensitivity (psychological) | Throughout study completion, on average 1 year
  Psychological stress sensitivity is measured through subjective stress reports of the participants using the visual analogue scale (VAS). VAS scorings are taken before, during, and after a stress task performed during the pre-intervention and post-intervention visit.
Fear (biological) | Throughout study completion, on average 1 year
  Fear-related processes will be explored using a computerized task. Biological fear response is measured using skin conductance, and a skin conductance response (μS) is calculated .
Fear (psychological) | Throughout study completion, on average 1 year
  Fear-related processes will be explored using a computerized task. Psychological fear response is measured subjectively by asking participants to indicate their expectancy score of an aversive stimulus.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | Throughout study completion, on average 1 year
  Assessing ratings on the subscales of PANAS, positive and negative affect, before and after intervention. PA subscale scores range between 10-50, with higher scores indicating better outcome. NA subscale scores range between 10-50, with higher scores indicating worse outcome.
Perceived Stress Scale (PSS) | Throughout study completion, on average 1 year
  Assessing ratings on PSS before and after intervention. PSS scores range between 0-40 with higher scores indicating worse outcome.
Gastrointestinal Symptom Rating Scale (GSRS) | Throughout study completion, on average 1 year
  Assessing ratings on the subscales of GSRS and its total score before and after intervention. It has 5 subscales (Reflux, Diarrhea, Constipation, Abdominal Pain, and Indigestion Syndrome). Subscale scores range from 1 to 7 and higher scores indicates a worse outcome.
Leiden Index of Depression Sensitivity (LEIDS-R) | Throughout study completion, on average 1 year
  Assessing ratings on the subscales of LEIDS-R and its total score before and after intervention. This is a self-report on cognitive reactivity comprised of 34 items with six subscales. Hopelessness/suicidality; Acceptance/Coping; Aggression; Control/Perfectionism; Risk Aversion; Rumination.
State-Trait Anxiety Inventory, State Anxiety Subscale (STAI-S) | Throughout study completion, on average 1 year
  Assessing ratings on the momentary (state) anxiety subscale of STAI before and after intervention. This is a self-report comprised of 20 questions specifically for state anxiety, rated on a 4-point scale. State anxiety is rated with anxiety absent and anxiety present questions. Anxiety absent questions constitute the absence of anxiety in a statement like, "I feel secure." Anxiety present questions represent the presence of anxiety in a statement like "I feel worried." The 4-point scale are as follows: 1 'not at all', 2 'somewhat', 3 'moderately so', and 4 'very much so'.
Brain response to stress | Throughout study completion, on average 1 year
  Brain response (brain oxygenation level-dependent signals) to a fMRI-adapted stress task will be measured before and after intervention

OTHER OUTCOMES:
Fecal gut microbiota profile | Throughout study completion, on average 1 year
  Assessing gut microbiota profile before and after intervention
Serum short-chain fatty acid levels | Throughout study completion, on average 1 year
  Quantification of serum SCFA (μM) before and after intervention
Cytokine levels | Throughout study completion, on average 1 year
  Quantification of inflammatory cytokines (pg/ml) before and after intervention
C-reactive protein levels | Throughout study completion, on average 1 year
  Quantification of C-reactive protein levels (ng/ml) before and after intervention
Heart rate variability | Throughout study completion, on average 1 year
  Assessing heart rate variability (ms) with ECG before and after intervention
Heart rate | Throughout study completion, on average 1 year
  Assessing heartbeat (bpm) with a blood pressure monitor before and after intervention
Blood pressure | Throughout study completion, on average 1 year
  Assessing blood pressure (systolic/diastolic mmHg) with a blood pressure monitor before and after intervention
Brain metabolite concentration | Throughout study completion, on average 1 year
  Relative quantification of brain metabolites (mmol/L) using 1H-Magnetic Resonance Spectroscopy before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, MD, PhD, Principal Investigator — KU Leuven; Kristin Verbeke, Pharm, PhD, Principal Investigator — KU Leuven; Boushra Dalile, PhD, Principal Investigator — KU Leuven; Jeroen Raes, PhD, Principal Investigator — VIB-KU Leuven
Locations (1):
- UZ/KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication will be made available to other researchers with all identifying information removed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available upon publication with no time limitations.
Access Criteria: The data will be publicly available.